CLINICAL TRIAL: NCT06955182
Title: Dynamic Hot Spring Hydrotherapy for Gait Disorders and Balance Function Recovery After Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Liqing Yao, Department of rehabilitation medicine, the Second Affiliated Hospital of Kunming Medical University, The Second Affiliated Hospital of Kunming Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shen-PJ-Ke-2025-19
Record Dates: First submitted 2025-04-14; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional rehabilitation intervention (Sham Comparator): Under closed management, patients will receive routine physical therapy for 40 minutes 5 times a week: 1) 20 minutes of routine rehabilitation, including routine muscle strength enhancement training, joint range of motion training, and neuropathological methods (Bobath method, proprioceptive neuromuscular facilitation technique, etc.); 2) 20 minute land balance walking function training
  Interventions: Other: Conventional rehabilitation intervention
- Dynamic hot spring hydrotherapy intervention (Experimental): Under closed management, patients will receive 5 times a week, 20 minutes of routine rehabilitation and 20 minutes of hot spring water exercise each time: (1) 20 minutes of routine rehabilitation: including routine muscle strength enhancement training, joint range of motion training, and neuropathological methods (Bobath method, proprioceptive neuromuscular facilitation technique, etc.); (2) 20 minute hot spring water balance walking function training
  Interventions: Other: Dynamic hot spring hydrotherapy intervention

INTERVENTIONS:
Other: Dynamic hot spring hydrotherapy intervention — Under closed management, patients will receive 5 times a week, 20 minutes of routine rehabilitation and 20 minutes of hot spring water exercise each time: (1) 20 minutes of routine rehabilitation: including routine muscle strength enhancement training, joint range of motion training, and neuropathological methods (Bobath method, proprioceptive neuromuscular facilitation technique, etc.); (2) 20 minute hot spring water balance walking function training
  Arms: Dynamic hot spring hydrotherapy intervention
Other: Conventional rehabilitation intervention — Under closed management, patients will receive routine physical therapy for 40 minutes 5 times a week: 1) 20 minutes of routine rehabilitation, including routine muscle strength enhancement training, joint range of motion training, and neuropathological methods (Bobath method, proprioceptive neuromuscular facilitation technique, etc.); 2) 20 minute land balance walking function training
  Arms: Conventional rehabilitation intervention

SUMMARY:
Our research aims to analyze and compare the improvement of various indicators of gait disorders and balance function before and after dynamic hot spring hydrotherapy and conventional exercise intervention, and clarify the therapeutic effect of dynamic hot spring hydrotherapy on gait disorders and balance function in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cerebral infarction or cerebral hemorrhage who meet the diagnostic criteria for stroke of the Chinese Medical Association; (2) Initial stroke<6 months, or last stroke event>6 months; (3) Age>=18 years old,<85 years old (increased risk of VCI over 85 years old); (4) NIHSS>4, NIHSS<26 points; (5) MRS score>=2 points; (6) complete CT or MRI; (7) No serious neurological or mental illness; Unconscious disorders, able to cooperate with relevant treatments; No severe cognitive impairment (MMSE>=15 points); (8) Berg Balance Scale>40 points; (9) The patient or family member signs an informed consent form.

Exclusion Criteria:

* (1) Concurrent major diseases, such as heart, lung, liver, kidney and other organ diseases or failure; (2) There are contraindications for hydrotherapy such as acute infectious diseases, open skin wounds, and severe epilepsy; (3) There are other clinical issues that may affect the assessment results, such as low vision, fractures, vestibular diseases, etc; (4) There are other neurological disorders, such as multiple sclerosis, Parkinson's disease, etc; (5) Serious mental and psychological problems exist; (6) Malignant tumor patients; (7) Early pregnancy or high-risk pregnancy; (8) Serious alcohol abusers; (9) Patients with active bleeding, such as gastrointestinal bleeding, nosebleeds, and excessive menstruation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go Test, (TUG) | From enrollment to the end of treatment at 2 weeks.
  Timed Stand Up Walking Test (TUG)
  Assess gait based on the time required for the test subject to stand up from the chair, walk at a steady pace to the 3-meter mark, and then return to the chair to sit down. The evaluation results are as follows:
  <10 seconds: Normal activity ability, low risk of falling. 10-14 seconds: There may be mild functional impairment, further evaluation is needed.
  >14 seconds: The risk of falling significantly increases (such as in elderly people or Parkinson's disease patients).
  >20 seconds: Prompt for severe mobility impairment, requiring intervention (such as in post-stroke patients).
10 Meter Walk Test, (10WMT) | From enrollment to the end of treatment at 2 weeks.
  Individuals walk 10 meters and have participants conduct 3 trials at a comfortable walking speed, followed by 3 trials at the patient's fast walking speed. Measure the middle 6 meters, allowing for acceleration and deceleration. The timing starts when the toe of the current foot crosses the 2-meter mark; The timer ends when the toe of the current foot crosses the 8-meter mark; In units of s, accurate to two decimal places; Calculate the average for each walking speed. The actual speed is 6m divided by the recorded seconds to obtain the speed in m/s. The speed rating results are as follows:
  <0.4m/s can be used for family walking 0.4-0.8m/s allows for limited community walking >0.8m/s can be used for community walking If the test subject requires full assistance, a score of 0 should be recorded.
Berg Balance Scale, BBS | From enrollment to the end of treatment at 2 weeks.
  The BBS consists of 14 projects, including sitting to stand, standing independently, sitting independently, standing to sit, bed chair transfer, standing with closed eyes, standing with both feet together, extending the upper limbs in the standing position, picking up objects from the ground in the standing position, turning around to look back, turning around once, alternating steps with both feet, standing on one leg, etc. Each project is rated from 0 to 4 points based on the patient's completion status, with a total score of 56 points. The evaluation results are as follows:
  41-56 points: Good balance function, low risk of falling 21-40 points: There is a certain degree of decline in balance function, and the risk of falling is moderate 0-20 points: Severe impairment of balance function, high risk of falling
Fugl-Meyer Balance Assessment,（FMA-B) | From enrollment to the end of treatment at 2 weeks.
  The ability of the test subject to complete various balance test items, including unsupported sitting; Healthy side "spreading wings" reaction; The completion of the "spreading wings" reaction on the affected side, standing with support, standing without support, standing on the healthy side, and standing on the affected side will be scored. Each examination item will be scored on a scale of 0-2 points, with the highest score of 14 points and the lowest score of 0 points. If the score is less than 14 points, it indicates that the balance function is impaired. The lower the score, the more severe the balance dysfunction.
Forced Vital Capacity, (FVC). | From enrollment to the end of treatment at 2 weeks.
  Typically, adult males consume 3000~5000ml, while females consume 2000~4000 liters.
FEV1 | From enrollment to the end of treatment at 2 weeks.
  The amount of gas exhaled in the first second is approximately 3179 ± 117mL for normal males and 2314 ± 48mL for females, starting from the maximum inhalation to the level of total lung volume.
Maximum Voluntary Ventilation, (MVV) | From enrollment to the end of treatment at 2 weeks.
  The general normal standard for pulmonary function MVV is: Male: （104+2.71)L/min； female sex: （82.5+2.17）L/min。
VO2 | From enrollment to the end of treatment at 2 weeks.
  The maximum amount of oxygen that the human body can absorb per unit time during exercise is usually measured in milliliters per minute (ml/min). VO2 reflects the cardiovascular function and aerobic exercise capacity of the human body, and is an important indicator for evaluating human endurance.
oxygen consumption per kg body weight, (VO2/Kg) | From enrollment to the end of treatment at 2 weeks.
  Oxygen consumption per unit weight (kg) per unit time. Expressed in VO2/kg. It is an indicator of an individual's athletic ability.The unit is mL/(kg · min).
METS | From enrollment to the end of treatment at 2 weeks.
  METs (metabolic equivalents) are indicators of energy expenditure during physical activity. 1 MET is equal to the oxygen consumption during sitting (approximately 3.5 mL/kg/min).
Respiratory Quotient, (RQ) | From enrollment to the end of treatment at 2 weeks.
  RQ refers to the ratio of carbon dioxide production to oxygen consumption in the body, and is commonly used to evaluate the energy metabolism of the body in different states. The numerical range of RQ is between 0.67 and 1.3.
VE | From enrollment to the end of treatment at 2 weeks.
  It is the amount of ventilation that maintains normal gas exchange in a resting state, equal to tidal volume multiplied by respiratory rate per minute.The unit is L/min.
breathing reserve ratio | From enrollment to the end of treatment at 2 weeks.
  BR=Maximum Ventilation Volume (MVV) - Minute Ventilation Volume during Maximum Exercise (VE).Normal respiratory reserve should be greater than 15L/min, indicating normal dynamic lung function levels in the body.
Tidal Volume, (VT) | From enrollment to the end of treatment at 2 weeks.
  VT is the amount of gas entering and leaving the lungs during each breath, reflecting the ventilation function of the lungs. The normal range for adults is about 6-8 milliliters per kilogram of body weight.
Heart Rate, (HR) | From enrollment to the end of treatment at 2 weeks.
  Heart rate is an important indicator of the human cardiovascular system, which reflects the functional status of the heart. HR can refer to instantaneous heart rate, measured in beats per minute.
VO2/WR | From enrollment to the end of treatment at 2 weeks.
  Under normal physiological conditions, there is a linear relationship between VO2 and the power of the human body to do work, commonly expressed as VO2/WR, with the unit of m/(min · W). The normal value is 8.4~11ml/(min · W). Decreased VO2/WR often indicates impaired oxygen delivery.
The oxygen pulse (VO2/HR) | From enrollment to the end of treatment at 2 weeks.
  The oxygen pulse is calculated by dividing VO2 by the heart rate at the same time. It is the amount of oxygen taken into the lung blood during one heart beat, which is equal to the product of the output per beat and the arterial mixed venous oxygen content difference [C (a-v) O2]. Its unit is ml/kg/min.
VO2@AT | From enrollment to the end of treatment at 2 weeks.
  It refers to the oxygen uptake at the anaerobic threshold (AT). The normal value of peakVO2 is usually greater than 40%, which is equivalent to 50%~65% peakVO2.
PetCO2 | From enrollment to the end of treatment at 2 weeks.
  It refers to the pressure value of carbon dioxide in the exhaled gas at the end of exhalation. By monitoring PetCO2, the condition of lung ventilation and blood flow can be reflected. The normal value of PetCO2 (end tidal carbon dioxide partial pressure) is 35-45 mmHg.
PetO2 | From enrollment to the end of treatment at 2 weeks.
  It reflects the oxygen partial pressure in the alveolar gas at the end of exhalation, and the normal range of PetO2 is 95-100mmHg
VE/VO2 | From enrollment to the end of treatment at 2 weeks.
  VE/VO2 refers to the ratio of minute ventilation to minute oxygen consumption, which is normally between 25-35.
VE/VCO2 | From enrollment to the end of treatment at 2 weeks.
  VE/VCO2 refers to the ratio of minute ventilation to minute carbon dioxide emissions, with a normal range of 30-40.
SpO2 | From enrollment to the end of treatment at 2 weeks.
  SpO2 refers to pulse oximetry, and the normal range of SpO ₂ for normal adults in a calm breathing state at sea level is 95% -100%.
HR_1_minute | From enrollment to the end of treatment at 2 weeks.
  It usually refers to the number of heartbeats counted within one minute, with a focus on specific heart rate values per minute. Under normal circumstances, the heart rate of adults in a quiet state is generally 60-100 beats per minute.
P Syst | From enrollment to the end of treatment at 2 weeks.
  It refers to the pressure exerted by blood on the walls of blood vessels during cardiac contraction, at which the ventricles pump blood into the aorta, causing the pressure inside the aorta to rise to its highest value, usually measured in mmHg (millimeter of mercury). The normal range of systolic blood pressure for normal adults in a quiet state is usually 90-139mmHg.
P Diast | From enrollment to the end of treatment at 2 weeks.
  It is the pressure exerted on the blood vessel walls during diastole, when the ventricles are in a filled state and the pressure inside the aorta drops to its lowest value. The normal range of diastolic blood pressure for normal adults in a quiet state is generally 60-89mmHg.
Step Length | From enrollment to the end of treatment at 2 weeks.
  The horizontal distance from the same foot following the ground to the opposite foot following the ground (left/right step lengths may be asymmetric).Its unit is meters.
Stride Length | From enrollment to the end of treatment at 2 weeks.
  The horizontal distance between two consecutive landings of the heel on the same side (one complete gait cycle).Its unit is meters.
Step Width | From enrollment to the end of treatment at 2 weeks.
  The lateral distance between the inner edges of both feet, reflecting walking stability.Its unit is meters.
Cadence | From enrollment to the end of treatment at 2 weeks.
  Steps per minute (steps/minute), typically around 100-120 steps for adults.
Walking Speed | From enrollment to the end of treatment at 2 weeks.
  The distance traveled per unit of time (in meters per second), which comprehensively reflects gait function.
Stance Phase | From enrollment to the end of treatment at 2 weeks.
  The proportion of time the foot is in contact with the ground (approximately 60% of the normal gait cycle).
Swing Phase | From enrollment to the end of treatment at 2 weeks.
  The proportion of time spent swinging the foot off the ground (usually around 40%).
Double Support | From enrollment to the end of treatment at 2 weeks.
  The time for both feet to touch the ground simultaneously (prolonged when the pace slows down).Its unit is seconds.
Hip joint | From enrollment to the end of treatment at 2 weeks.
  Sagittal flexion/extension (normal range of approximately 30 ° flexion to 10 ° extension).
Knee joint | From enrollment to the end of treatment at 2 weeks.
  Sagittal plane flexion (0 ° extension to 60 ° flexion swing phase).
Ankle joint | From enrollment to the end of treatment at 2 weeks.
  Sagittal dorsiflexion/plantarflexion (dorsiflexion when the foot touches the ground, plantarflexion during advancement).
Pelvic movements | From enrollment to the end of treatment at 2 weeks.
  Forward/backward tilt, internal and external rotation, lateral tilt.
Ground Reaction Force (GRF) | From enrollment to the end of treatment at 2 weeks.
  Measured by a force measuring platform, a typical bimodal curve (first peak ≈ 110% of body weight, second peak ≈ 120% of body weight).
Joint Moments | From enrollment to the end of treatment at 2 weeks.
  Reflecting the control of muscles and ligaments over joints (such as predicting the risk of osteoarthritis with knee adduction torque).The unit of it is N · m (Newton meters)
Power | From enrollment to the end of treatment at 2 weeks.
  Joint work efficiency (peak power during ankle joint propulsion is key).The unit it is W.
Symmetry Index | From enrollment to the end of treatment at 2 weeks.
  The difference in step size and support phase time between the left and right sides (often asymmetric in stroke patients).
Phase Coordination | From enrollment to the end of treatment at 2 weeks.
  The temporal relationship between the swing phase and the support phase (which may be disrupted in Parkinson's disease patients).
Center of gravity position | From enrollment to the end of treatment at 2 weeks.
  It refers to the projection position of the center of gravity on the horizontal plane when the human body is standing quietly. By using pressure tablets and other devices, the front, back, left, and right positions of the center of gravity can be measured, reflecting the body's balance state under static conditions. Under normal circumstances, the center of gravity is relatively stable and within the range of the area supported by both feet.
Center of gravity swing amplitude | From enrollment to the end of treatment at 2 weeks.
  It refers to the maximum distance that the center of gravity deviates from the center position within a certain period of time. The smaller the swing amplitude, the better the static balance ability. Generally measured in millimeters (mm), when healthy adults stand quietly, the amplitude of their center of gravity swing back and forth is usually around 10-20mm, and the amplitude of left and right swing is relatively small.
Center of gravity swing frequency | From enrollment to the end of treatment at 2 weeks.
  It refers to the number of times the center of gravity swings per unit time. The lower the frequency, the stronger the static balance control capability. When a normal adult stands quietly, the frequency of center of gravity swing is generally between 0.5-2 times per second.
Walking stability | From enrollment to the end of treatment at 2 weeks.
  It is evaluated by analyzing the step characteristics during walking, including step length, stride length, step frequency, bipedal support time, single foot support time, and other parameters. For example, if the stride is uniform, the stride is stable, the stride frequency is moderate, and the ratio of foot support time to single foot support time is reasonable, it indicates good dynamic balance ability during walking. When adults walk normally, the stride length is about 50-80cm, and the step frequency is around 90-120 steps per minute.
Posture transition ability | From enrollment to the end of treatment at 2 weeks.
  It measures the stability and coordination during the transition from one posture to another (such as sitting to standing, standing to walking, etc.). The evaluation indicators include conversion time, accuracy of center of gravity shift, and whether additional support or auxiliary movements are needed. Healthy individuals complete posture transitions quickly and smoothly, with a smooth shift of center of gravity, typically without the need for external force or excessive adjustment movements.
Disturbance response ability | From enrollment to the end of treatment at 2 weeks.
  The ability of the human body to restore balance through its own balance adjustment mechanism when subjected to external disturbances such as sudden thrust, tension, or ground shaking. The relevant parameters include reaction time, maximum offset distance, and time to restore balance. Rapid response, ability to control the body's center of gravity within a small deviation range and quickly restore balance, indicate good disturbance response ability.
Visual dependence level | From enrollment to the end of treatment at 2 weeks.
  It is evaluated by comparing the balance test results between open and closed eye states. If the balance function significantly decreases after closing the eyes, it indicates a high degree of dependence on visual information; On the contrary, if there is not much difference in balance performance between opening and closing the eyes, it indicates that other balance regulation mechanisms such as proprioception have played a good role. For example, in the test of standing on one foot with closed eyes, the ability to stand for a longer period of time when the eyes are open is significantly reduced, indicating that vision plays an important role in maintaining balance in this posture.
Muscle activity pattern | From enrollment to the end of treatment at 2 weeks.
  Using techniques such as surface electromyography to record the activation sequence, intensity, and duration of different muscles during balance tasks. Normal balance control requires multiple groups of muscles to work together, and whether the muscle activity pattern is normal or not can reflect the nervous system's ability to control muscles and the coordination and cooperation between muscles. For example, when maintaining balance in a standing position, the calf muscles, hip muscles, and back muscles will contract and relax in a timely manner according to changes in the body's center of gravity to maintain stability.

SECONDARY OUTCOMES:
anxiety | From enrollment to the end of treatment at 2 weeks
  Beck Anxiety Inventory Scoring is based on the severity of anxiety symptoms, and the total score is calculated by adding up each result. Scores 15-25 indicate mild anxiety, 26-35 indicate moderate anxiety, and scores above 36 indicate severe anxiety.
sleep quality | From enrollment to the end of treatment at 2 weeks
  Pittsburgh Sleep Quality Index (PSQI) According to the various indicators of sleep quality, the frequency is divided into 0-5 points: good sleep quality, 6-10 points: decent sleep quality, 11-15 points: average sleep quality, 16-21 points: poor sleep quality.
Self efficacy | From enrollment to the end of treatment at 2 weeks
  ABC Balanced Confidence Scale Based on the confidence level of each item, ranging from 0% (no confidence) to 100% (completely confident), the total score is taken as the average of all items.
  ≥ 80%: Good balance and confidence, low risk of falling; 50%~80%: moderate risk; <50%: High risk, requiring intervention.
Neurotransmitters and Cytokines | From enrollment to the end of treatment at 2 weeks
  β - endorphin, tumor necrosis factor - α (TNF - α), and interleukin-6 (IL-6)

CONTACTS AND LOCATIONS:
Locations (1):
- Electroencephalography, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Undecided